CLINICAL TRIAL: NCT05151887
Title: The Impact of Ingesting a Whole-food Animal-based Versus Plant-based Protein Rich Meal on the Muscle Protein Synthetic Response in Healthy Older Men and Women
Brief Title: The Impact of a Whole-food Animal-based Versus Plant-based Protein Rich Meal on Muscle Protein Synthesis
Acronym: MeaL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry); Vion Food Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: METC 21-006
Record Dates: First submitted 2021-11-15; First posted 2021-12-09 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Muscle Protein Synthesis; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: The present study utilizes a randomized, counter-balanced, cross-over design in healthy older male and female participants. In total, 16 healthy older men and women (1:1 ratio of men:women) will participate in the study (20 including potential drop-out). Participants will be randomly assigned to either receive the meal including meat or exclusively plant based foods during the Test Day 1. During Test Day 2, participants will receive the other meal.
Masking Description: In this trial, neither the participants, nor the researchers who perform the trial days will be blinded to the intervention allocation. However, the researchers performing the sample analysis are blinded to intervention allocation and are not involved in the research study during the trial days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meat meal (Experimental): Minced beef, potato, string beans, apple sauce, and herb butter
  Interventions: Other: Muscle protein synthesis
- Plant meal (Experimental): Quinoa, soy beans, chickpeas, broad beans, and soy sauce
  Interventions: Other: Muscle protein synthesis

INTERVENTIONS:
Other: Muscle protein synthesis — The meals contain a total of 0.45 g protein/kg body mass (36 g protein for an 80 kg person). To account for differences in body mass, the investigators will scale the meal content to ensure 0.45 g/kg body mass for different body mass ranges (i.e., 65-75 kg, 75-85 kg, etc.). As such, carbohydrate, fat, and total energy content of the meals will also be scaled to body mass. The test meals are composed out of regular whole food items which will be purchased from local shops. The muscle protein synthetic response following meal ingestion will be assessed by the use of stable isotope tracer methodology

SUMMARY:
Rationale: Food intake stimulates muscle protein synthesis rates. The magnitude of the anabolic response to feeding forms a key factor in regulating muscle mass maintenance. Ingestion of animal-derived proteins generally leads to a greater stimulation of muscle protein synthesis when compared to the ingestion of plant-derived proteins. What is often neglected is that the anabolic properties of protein isolates do not necessarily reflect the anabolic response to the ingestion of the whole-foods from which those are derived. This discrepancy is due to the presence or absence of other components normally found within whole-food matrices, which influence protein digestion and amino acid absorption from animal based and plant based protein sources. A rapid and robust post-prandial release of food-derived amino acids is of particular relevance for older individuals, who typically show a blunted muscle protein synthetic response to feeding

Objective: To compare the post-prandial muscle protein synthetic response following ingestion of a whole-food meal (560 kilo calorie (kCal); ~36 g protein total, ~0.45 g/kg body weight) containing ~100 g lean ground beef (~30 g protein) versus the ingestion of an isonitrogenous, isocaloric whole-food meal containing only plant-based protein sources (561 kCal; ~36 g protein total) in vivo in healthy, older men and women.

Study design: randomized, counter-balanced, cross-over design, researchers and participants are not blinded, analysts are blinded.

Study population: 16 healthy older (65-85 y) men and women (1:1 ratio of men:women)

Intervention: Participants will undergo 2 test days. On one test day participants will consume a whole-food meal containing meat as the primary source of protein (~36 g, ~0.45 g/kg body weight). On the other day, participants will consume a whole-food meal containing only plant-based foods as the source of protein (~36 g or ~0.45 g/kg body weight). In addition, a continuous intravenous tracer infusion will be applied, and blood an muscle samples will be collected in order to assess the muscle protein synthetic response.

Main study parameters/endpoints: The primary endpoint will be mixed muscle protein synthesis rates over the full 6h post-prandial period following meal ingestion.

DETAILED DESCRIPTION:
Food intake stimulates muscle protein synthesis rates. The anabolic response to feeding forms a key factor in regulating muscle mass maintenance. Impairments in the sensitivity of skeletal muscle tissue to respond to the anabolic properties of protein feeding have been reported in numerous settings where muscle mass is being lost, such as aging, disuse, chronic metabolic disease, and various clinical conditions where muscle wasting is apparent.

The capacity of a dietary protein to stimulate post-prandial muscle protein accretion depends on the digestion and absorption kinetics of that protein as well as its amino acid composition. A more rapid rise in circulating essential amino acids (EAAs), with leucine in particular, drives the post-prandial rise in muscle protein synthesis rates. It has been suggested that plant and animal based protein sources do not have the same anabolic properties due to differences digestibility and essential amino acid composition. However, so far, nearly all studies evaluating the muscle protein synthetic response to food ingestion have applied a reductionist approach and have determined the muscle protein synthetic response to the ingestion of isolated protein sources (e.g., whey, casein, soy) with or without other isolated meal components (e.g., carbohydrates, fats). This work suggests that the ingestion of isolated animal-based proteins stimulates a superior muscle protein synthetic response when compared to the ingestion of isolated plant-based proteins. However, protein isolates never constitute the main protein portion of a meal. Perhaps more importantly, it is often neglected that the anabolic properties of protein isolates do not necessarily reflect the anabolic response to the ingestion of the whole-foods from which those are derived. This discrepancy is due to the presence or absence of other nutritional components within whole-food matrices. In particular, plant-derived protein sources contain anti-nutritional factors that impair protein digestion and amino acid absorption and, as such, compromise the post-prandial rise in muscle protein synthesis rates.

Therefore, this project will compare the impact of the ingestion of a whole-food meal with beef as the primary source of protein, with the ingestion of a whole food meal ingestion with only plant derived protein sources, on the muscle protein synthetic response in healthy older men and women.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-85 years
* Body mass index 18.5 - 30 kg/m2
* Healthy
* Having given informed consent

Exclusion Criteria:

* Allergy for one of the food items used
* >5% weight change in the previous 6 months
* Participating in a structured (progressive) exercise program
* Smoking
* Diagnosed musculoskeletal disorders
* Diagnosed metabolic disorders (e.g. diabetes)
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories).
* Chronic use of gastric acid suppressing medication
* Chronic use of anti-coagulants
* Diagnosed GI tract disorders or diseases
* Blood donation in the past 2 months
* Strict vegetarian diet

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis rates | One integrative value over the 6 hour post-prandial period
  Post-prandial muscle protein synthesis rates Meat meal vs Plant meal

SECONDARY OUTCOMES:
Muscle protein synthesis rates | -3-0 hour, 0-3 hour, and 3-6 hour
  Muscle protein synthesis rates during the basal period and over 0-3 hour and 3-6 hour period
Plasma amino acid concentrations | 6 hour post-prandial period
  Post-prandial plasma amino acid availability
Plasma glucose concentrations | 6 hour post-prandial period
  Post-prandial plasma glucose availability
Plasma insulin concentrations | 6 hour post-prandial period
  Post-prandial plasma insulin availability

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinckaers PJ, Domic J, Petrick HL, Holwerda AM, Trommelen J, Hendriks FK, Houben LH, Goessens JP, van Kranenburg JM, Senden JM, de Groot LC, Verdijk LB, Snijders T, van Loon LJ. Higher Muscle Protein Synthesis Rates Following Ingestion of an Omnivorous Meal Compared with an Isocaloric and Isonitrogenous Vegan Meal in Healthy, Older Adults. J Nutr. 2024 Jul;154(7):2120-2132. doi: 10.1016/j.tjnut.2023.11.004. Epub 2023 Nov 15. PMID 37972895